CLINICAL TRIAL: NCT05157217
Title: Impact of the Genetic Polymorphism on the Severity of COVID-19 Infection in Egyptian Patients
Brief Title: Impact of the Genetic Polymorphism on COVID-19 in Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Naglaa Samir Ahmed Bazan, Ass. Professor and Acting Head of Clinical Pharmacy Department - Cairo University Hospitals, Cairo University
Other Study IDs: N-134-2020
Record Dates: First submitted 2021-12-11; First posted 2021-12-14 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: COVID-19; Genetic Polymorphism; Pharmacogenetics
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A baseline blood sample 3 ml on EDTA tube for genotyping of the studied alleles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: COVID-19 carriers who were infected with SARS-CoV-2 and healed without suffering from any respiratory complications or the need for hospitalization
- Group 2: COVID-19 patients who suffered from serious respiratory complications that needed hospitalization or admission to the ICU

SUMMARY:
The COVID-19 infection severity depends on many factors, including genetic factors. The SNPs of ACE1, ACE2 and TMPRSS2; which have a big role in the viral entry to the cells, will be tested and help establish a relationship between the genetic variation in these SNPs and the severity of the COVID-19 symptoms. The aim of this study is to detect the association between ACE1, ACE2 and TMPRSS2 gene polymorphism variants and occurrences of severe complications in Egyptians patients with COVID-19 disease.

DETAILED DESCRIPTION:
The world has been battling with the COVID-19 pandemic since the end of 2019, which is caused by the highly contagious SARS-CoV-2 with over 25 million confirmed cases all around the world. Although it has been the focus of many studies, this new pandemic is still an enigma in many ways. The severity of the symptoms can vary from mild symptoms with flu-like symptoms and self-limiting disease to severe respiratory symptoms that needs hospitalization and ICU admission and can lead to death. Several factors have been speculated to affect the severity of the COVID-19 infection including genetic factors. In this study, we will investigate the variation in three different SNPs, one for the ACE2 gene which is the binding receptor for the SARS-CoV-2 virus (rs908004, consequence: 3 Prime UTR Variant, Alleles: C>G / C>T), one for the ACE (I/D) gene; which can in term affect the ACE2 receptor and the probability for lung injury ( rs4343, Consequence: Synonymous Variant, Alleles: G>A), and one for the TMPRSS2 gene; which is a transmembrane protease which activates the viral spike by priming it when it is attached to the ACE2 receptor ( rs12329760, consequence: Missense Variant, Alleles: C>T), and conclude if they have any effect in the COVID-19 disease severity and need for hospitalization and admission to the ICU. The aim is:

* To detect the incidence of angiotensin-converting enzyme Insertion/Deletion (ACE I/D), angiotensin-converting enzyme 2 (ACE2) and type 2 transmembrane serine protease (TMPRSS2) gene polymorphisms in the Egyptian population.
* To detect association between angiotensin-converting enzyme Insertion/Deletion (ACE I/D) gene polymorphism variants and occurrences of severe complications in patients with COVID-19 disease.
* To detect association between angiotensin-converting enzyme 2 (ACE2) gene polymorphism variants and occurrences of severe complications in patients with COVID-19 disease.
* To detect association between type 2 transmembrane serine protease (TMPRSS2) gene polymorphism variants and occurrences of severe complications in patients with COVID-19 disease.
* To investigate the potential interaction between ACE (I/D), ACE2 and TMPRSS2 gene polymorphisms and the occurrences of severe complications in patients with COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

Ø Positive nasal Swap for COVID-19 Infection. Ø Age of 18 years to 80 years. Ø Written informed consent of the subject to participate in the study.

Exclusion Criteria:

Ø Patients with any prior respiratory problems such Asthma and COPD.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Egyptian patients who are either : infected with SARS-CoV-2 and healed without suffering from any respiratory complications or the need for hospitalization Or infected with SARS-CoV-2 who suffered from serious respiratory complications that needed hospitalization or admission to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
ACE I/D gene polymorphism (rs4343) | 3 months
  Genotypic and allele frequencies of the studied SNPS in both study groups
Angiotensin-converting enzyme 2 (ACE2) gene polymorphism (rs908004) | 3 months
  Genotypic and allele frequencies of the studied SNPS in both study groups
Type 2 transmembrane serine protease (TMPRSS2) gene polymorphism (rs12329760) | 3 months
  Genotypic and allele frequencies of the studied SNPS in both study groups

SECONDARY OUTCOMES:
Potential interaction between ACE (I/D), ACE2 and TMPRSS2 gene polymorphisms and the occurrences of severe complications in patients with COVID-19 disease.1 | 3 months
  Genotypic and allele frequencies of all studied SNPS in patients who suffered from serious respiratory complications that needed hospitalization or admission to the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa S Bazan, PhD, Principal Investigator — Cairo University; Khaled Farouk, MD, Principal Investigator — Cairo University; Adel RA Abdallah, PhD, Study Chair — Al-Azhar University in Cairo; Abdelrahman A Abdelgawad, BScPharm, Principal Investigator — Misr International University; Neven MA Sarhan, PhD, Study Director — Misr International University; Raed SA Ismail, PhD, Study Director — Al-Azhar University in Cairo; Mohamed GL El-Ansary, MD, Study Director — Cairo University; Mona Schaalan, PhD, Study Director — Misr International University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol

REFERENCES:
- [Result] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Result] Zheng H, Cao JJ. Angiotensin-Converting Enzyme Gene Polymorphism and Severe Lung Injury in Patients with Coronavirus Disease 2019. Am J Pathol. 2020 Oct;190(10):2013-2017. doi: 10.1016/j.ajpath.2020.07.009. Epub 2020 Jul 29. PMID 32735889
- [Result] Asselta R, Paraboschi EM, Mantovani A, Duga S. ACE2 and TMPRSS2 variants and expression as candidates to sex and country differences in COVID-19 severity in Italy. Aging (Albany NY). 2020 Jun 5;12(11):10087-10098. doi: 10.18632/aging.103415. Epub 2020 Jun 5. PMID 32501810
- [Result] Hou Y, Zhao J, Martin W, Kallianpur A, Chung MK, Jehi L, Sharifi N, Erzurum S, Eng C, Cheng F. New insights into genetic susceptibility of COVID-19: an ACE2 and TMPRSS2 polymorphism analysis. BMC Med. 2020 Jul 15;18(1):216. doi: 10.1186/s12916-020-01673-z. PMID 32664879
- [Result] Itoyama S, Keicho N, Quy T, Phi NC, Long HT, Ha LD, Ban VV, Ohashi J, Hijikata M, Matsushita I, Kawana A, Yanai H, Kirikae T, Kuratsuji T, Sasazuki T. ACE1 polymorphism and progression of SARS. Biochem Biophys Res Commun. 2004 Oct 22;323(3):1124-9. doi: 10.1016/j.bbrc.2004.08.208. PMID 15381116